CLINICAL TRIAL: NCT05810389
Title: EVALUATION OF AN ALTERNATIVE TECHNIQUE FOR THE APPLICATION OF SODIUM FLUOROPHOSPHATE: A 2-YEARS DOUBLE-BLIND RCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Buenos Aires (Other)
Responsible Party: Principal Investigator, ALDO SQUASSI, Chairman Dept. Preventive and Community Dentistry, University of Buenos Aires
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IISAP-OPYC001
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Caries,Dental
MeSH Terms: conditions — Dental Caries | interventions — Fluorides

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- FFA toothbrush (Experimental)
  Interventions: Combination Product: Fluoride
- Varnish (Active Comparator)
  Interventions: Combination Product: Fluoride
- FFA gel (Active Comparator)
  Interventions: Combination Product: Fluoride

INTERVENTIONS:
Combination Product: Fluoride — Application methods of delivery of topical fluoride
  Other Names: Toothbrush

SUMMARY:
he study was designed as a double-blind three-parallel-group randomized controlled trial, in which the evaluators and a researcher, not involved in the evaluation process, was responsible for the randomization process, were masked to the group assignment.

The study will be carried out at 2 schools of the Metropolitan Area of Buenos Aires where school programs are developed by the Department of Preventive and Community Dentistry of the University of Buenos Aires, and that present homogeneous characteristics in terms of social risk. The children (n=244) attending those primary schools will be the population object of the trial.

Clinical examinations

Each child will go under a clinical examination to determine dental status according to the ICDAS II criteria (Pitts, 2005) and the Caries Treatment Need Index (CTNI).

Intervention

Children will be divided into three different groups according to the mode of treatment:

* NaF varnish group (NaFV) Professional application of 5% NaF varnish twice a year pH 7 (ClinPro White Varnish®) according to manufacturer's instructions.
* APF in tray Group (APFt) Professional application of APF 1.23% twice a year pH 3.5 (Klepp®) with tray according to manufacturer's instructions
* APF in toothbrush group (APFtbru) Professional application of APF 1.23% twice a year pH 3.5 (Klepp®) with toothbrush 2 minutes brushing according to manufacturer's instructions.

Dental examination and Monitoring

Observations and clinical examinations will be conducted at schools. After 12 and 24 months, the clinical examination will be repeated to assess the dental status of schoolchildren following the same criteria described. The presence of new caries lesions will be taken as a dependent variable. So sound surfaces on baseline will be observed for 24 months.

DETAILED DESCRIPTION:
The study was designed as a double-blind three-parallel-group randomized controlled trial, in which the evaluators and a researcher, not involved in the evaluation process, was responsible for the randomization process, were masked to the group assignment.

The study will be carried out at 2 schools of the Metropolitan Area of Buenos Aires where school programs are developed by the Department of Preventive and Community Dentistry of the University of Buenos Aires, and that present homogeneous characteristics in terms of social risk. The children (n=244) attending those primary schools will be the population object of the trial.

All parents/caregivers of the children will receive a leaflet requesting the approval to enroll their children; for those families that decide not to be included into the trial, the children will receive the dental treatment needed but their data will not be evaluated.

The inclusion criteria were children between 4 and 11 years old attending the selected schools. Exclusion criteria: Children with systemic diseases or systemic disease treatments, motor disorders and children receiving preventive measures in other public, private, or social security dental services.

Clinical examinations

Each child will go under a clinical examination to determine dental status according to the ICDAS II criteria (Pitts, 2005), perform under standardized conditions, using light, dental mirror, WHO probe and magnification (2,5x). The dental exams will be performed by calibrated researchers.

On the basis of the clinical examination, beside the ICDAS11,12 score, the Caries Treatment Need Index13 (CTNI) will also be registered.

Intervention

As described above, the children will be divided into three different groups according to the mode of treatment:

* NaF varnish group (NaFV) n=60 children Professional application of 5% NaF varnish twice a year pH 7 (ClinPro White Varnish®) according to manufacturer's instructions.
* APF in tray Group (APFt) n=60 children Professional application of APF 1.23% twice a year pH 3.5 (Klepp®) with tray according to manufacturer's instructions
* APF in toothbrush group (APFtbru) n=60 children Professional application of APF 1.23% twice a year pH 3.5 (Klepp®) with toothbrush 2 minutes brushing according to manufacturer's instructions.

Enrolment in each group will be given by balancing the CNTI categories in each group.

A protocol will be applied to all children, based on dental care programmes to be carried out in school and dental clinics, with the aim of controlling caries lesions, comprising: teaching and control of personal oral hygiene; dietary counseling, calculus removal, and caries treatment if needed.

Dental examination and Monitoring

Observations and clinical examinations will be conducted at schools. After 12 and 24 months, the clinical examination will be repeated to assess the dental status of schoolchildren following the same criteria described. The presence of new caries lesions will be taken as a dependent variable. So sound surfaces on baseline will be observed for 24 months.

In all children, daily brushing will be performed with the same toothpaste and toothbrush, supervised by schoolteachers, with fluoride toothpaste (1400 ppm) at school.

Statistical analysis

All the data will be input into a spreadsheet (Microsoft Excel 2021 for Mac, version 16.4.8). Chi -square test for NTCI changes between groups and after 24 months.

Kaplan - Meyer Statistical analyses will be performed using Stata/SE1 software, version Stata/SE 16.1 for Mac (Intel 64-bit)and SPSS 28 for survival of sound surfaces after 24 months and Hazard Ratio will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Schoolchildren

Exclusion Criteria:

-

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Caries incidence reduction | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: ALDO SQUASSI, Study Director — University of Buenos Aires
Locations (1):
- Universidad de Buenos Aires, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet